CLINICAL TRIAL: NCT03666728
Title: An Open-label, Single-arm, Multi-center, Phase 2 Study to Evaluate SHR-1210 Combination With BP102 in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer Whose PD-L1 Positive and EGFR/ALK Wild Type.
Brief Title: A Study of SHR-1210 in Combination With BP102 in Subjects With Non-squamous NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: changes in the R&D strategy
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-211
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+BP102 (Experimental): Subjects receive SHR-1210 200 mg and BP102 15 mg/kg in day 1 intravenously every 3 weeks, until disease progression or unacceptable toxicity.
  Interventions: Drug: SHR-1210; Drug: BP102

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 was administered 200 mg iv every 3 weeks
Drug: BP102 — BP102 was administered 15 mg/kg iv every 3 weeks

SUMMARY:
SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody. This is a Phase II, multicenter, open-label study designed to evaluate the safety and efficacy of SHR-1210 with BP102 in subjects who are chemotherapy naive and have Stage IIIB~IV non-squamous NSCLC. The primary end points are ORR and PFS.

In this study, subjects will receive SHR-1210 combined with BP102 until progression or unacceptable toxicity (SHR-1210 or BP102 for a maximum of 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1;
* Subjects who are chemotherapy naive and have Stage IIIB-IV non-squamous NSCLC;
* Gene diagnostic tests must show that subjects are with wild type of EGFR, ALK and ROS1;
* Known PD-L1 status as determined by immunohistochemistry assay performed on previously obtained archival tumor tissue or tissue obtained from a biopsy at screening;
* No prior systemic treatment;
* Adequate hematologic and end organ function;
* Female participants of childbearing potential must have a negative serum pregnancy test within -7 days of randomization and must be willing to use very efficient barrier methods of contraception or a barrier method plus a hormonal method starting with the screening visit through 6 months after the last dose Male participants with a female partner(s) of child-bearing potential must be willing to use very efficient barrier methods of contraception from screening through 6 months after the last dose.

Exclusion Criteria:

* Significant cardiovascular disease;
* Prior treatment with immune checkpoint blockade therapies, anti-programmed death-1, and anti-PD-L1 therapeutic antibodies;
* History of autoimmune disease;
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome;
* Severe infection within 4 weeks prior to randomization;
* Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation that such a live attenuated vaccine will be required during the study;
* Major surgical procedure within 4 weeks prior to randomization;
* History of hemoptysis within 12 weeks prior to randomization;
* Inadequately controlled hypertension;
* Evidence of bleeding diathesis or coagulopathy;
* Prior allogeneic bone marrow transplantation or solid organ transplant;
* Positive test for HIV, and patients with active hepatitis B or hepatitis C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 1 year
  ORR, determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Progression-Free Survival (PFS) | up to approximately 1 year
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment.

SECONDARY OUTCOMES:
Time to Response (TTR) | up to approximately 1 year
  Determined using RECIST v1.1 criteria
Duration of Response Rate (DoR) | up to approximately 1 year
  Determined using RECIST v1.1 criteria
Disease Control Rate (DCR) | up to approximately 1 year
  Determined using RECIST v1.1 criteria
Overall Survival Rate at 12-month (OSR) | up to 1 year
Number of participants with treatment-related adverse events (AEs) | up to approximately 1 year
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangsu HengRui Medicine Co., Ltd., Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China